CLINICAL TRIAL: NCT05292690
Title: An Assistive Powered Wheelchair: Stage 2 Trial - Powered Wheelchair User Evaluation of an Obstacle Alerting System. A Non-interventional Study
Brief Title: An Assistive Powered Wheelchair: Stage 2 Trial
Acronym: EDUCAT
Status: Completed | Type: Observational
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: University of Kent (Other); Sussex Community NHS Foundation Trust (Other); KU Leuven (Other); l'Institut supérieur de l'électronique et du numérique (ISEN) Lille (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020/MEDPHYS/01
Record Dates: First submitted 2022-02-02; First posted 2022-03-23 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis; Stroke; Cystic Fibrosis; Motor Neurone Disease; Craniocerebral Trauma; Guillain-Barre Syndrome
MeSH Terms: conditions — Multiple Sclerosis; Stroke; Cystic Fibrosis; Amyotrophic Lateral Sclerosis; Craniocerebral Trauma; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Powered Wheelchair Obstacle Alerting System — Evaluation of an Obstacle Alerting System

SUMMARY:
Preliminary evaluation of an obstacle alerting system to enhance the user's independent mobility by improving their confidence to drive and their safety in driving a powered wheelchair.

DETAILED DESCRIPTION:
Many powered wheelchair users find that collision free driving presents a significant challenge to confident and safe driving. In some cases so much so that the user will not drive their chair in some environments.

Interviews with users in the EDUCAT project confirmed that users had problems driving safely and confidently in a confined space, passing through doorways or down narrow corridors and when reversing.

Therefore the goal of this stage of the project is to improve the quality of life of the powered chair user by developing an obstacle alerting system which will help improve their confidence and safety in driving.

This was to be achieved by asking expert users to provide feedback on the impact and usefulness of providing information about the presence and location of obstacles in the vicinity of their powered wheelchair.

There are two aspects to this.

1. User assessment of the usefulness of the obstacle alerting feedback. This will include user evaluation of the value of the different modes of feedback - audio, visual and haptic - and how best to adapt these to the range of driving environments and driving speeds. And what level of control the user requires to select and deselect these options.
2. Monitoring the user's driving patterns with and without obstacle alerting -using the Stage 1 recording device.

The analysis of this data, and feedback from the Users and carers will inform the development and design of the obstacle alerting system.

Because of the COVID-19 pandemic the trial could not be carried out with powered wheel-chair users participating as they represented a clinically vulnerable part of the population. The trial was, therefore, adapted and carried out with adult non-wheelchair users.

ELIGIBILITY:
Inclusion Criteria:

1. Adults who are not wheelchair users.
2. Willing and able to provide a valid consent.
3. Able to participate in interviews aided or unaided using preferred method of communication.
4. Willing to drive a powered chair.

Exclusion Criteria:

1. Lacks capacity to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult non-powered wheelchair users
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Pre-trial Participant Evaluation of the possible Value of an Obstacle Alerting System | immediately before the intervention/procedure
  The participant had been given an information sheet describing the Obstacle Alerting System.
  The participants were given the pre-trial questionnaire to obtain their opinion of the value of the Obstacle Alerting System.
  In a face to face interview the participants were asked to score each question. 0=don't know, 1=not at all, to 5=very helpful. Participants were also asked to discuss the reasons for their choices.
  Questions included. Value of warning of obstacles in the vicinity of the powered chair. Use of visual, auditory and haptic feedback in a range of environments e.g. small room, lifts, corridor, doorways, crowded spaces.
  The value of a reversing camera.
  Perceived benefit for Powered Chair Users.
Post-trial Participant Evaluation of the possible Value of the Obstacle Alerting System | immediately after the intervention/procedure
  Post-trial questionnaire based on pre-trial questionnaire. Participants reassessed the Obstacle Alerting System [OAS] in the light of experience.
  In a face to face interview the participants were asked to score each question. 0=don't know, 1=not at all, to 5=very helpful. Participants were also asked to discuss the reasons for their choices.
  Asked when they found the OAS helpful and when unhelpful. Assessment of the feedback options and when they were and were not helpful. How could the OAS be improved to make it more user friendly and environment specific.
  Perceived benefit for Powered Chair Users.
Joystick range of movement patterns with and without the Obstacle alerting System Active | immediately after the intervention/procedure
  Range of movement scatter plots/ heat maps
Smoothness of joystick movement with and without the Obstacle alerting System Active | immediately after the intervention/procedure
  Smoothness of movement e.g. Normalised Jerk Score. A lower score indicates smoother and more controlled movements.
  Typical values for this trial are in the range of 3000-5000. A lower score is an indication of the participant learning to drive and becoming more familiar with the course.
  A lower score may occur with the Obstacle Alerting system active - if it helps. A higher score if it distracts. At present this is a novel measure of these factors
Joystick path length with and without the Obstacle alerting System Active | immediately after the intervention/procedure
  Joystick path length - distance the participant moves the joystick to drive the course. Calculated from the joystick displacement X and Y coordinates.
  For a set course it would be expected that the path length will decrease as the participant learns to drive and familiarises with the course. Fatigue not having an impact.
  A lower score may occur with the Obstacle Alerting system active - if it helps. A higher score if it distracts. At present this is a novel measure of these factors
Time to complete the course with and without the Obstacle alerting System Active | immediately after the intervention/procedure
  Manually timed. Start when participant enters the course, stop when exiting the course

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sakel, MD, Principal Investigator — East Kent Hospitals University Foundation Trust
Locations (1):
- East Kent Hospitals NHS Foundation Trust, Canterbury, Kent, United Kingdom

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT05292690/Prot_000.pdf
  • Study Protocol and Informed Consent Form: Informed Consent for Photographic Images (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT05292690/Prot_ICF_001.pdf
  • Informed Consent Form: Informed Consent to Participate in Trial (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT05292690/ICF_002.pdf